CLINICAL TRIAL: NCT00802867
Title: Safety and Immunogenicity of DAPTACEL® (CP10/5/5/3DT Aventis Pasteur 5-component Pertussis Vaccine in Combination With Tetanus and Diphtheria Toxoids Adsorbed) Administered as a 5th Dose in 4 to 6-Year-Old Children Previously Immunized With PENTACEL™ (HCP20/20/5/3DT-mIPV//PRP-T)
Brief Title: Study of DAPTACEL® Administered as a 5th Dose in 4 to 6-Year-Old Children Previously Immunized With PENTACEL™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P3T10
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2010-01-12 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Polio; Haemophilus Infection
Keywords: DAPTACEL®; PENTACEL™; Diphtheria; Tetanus; Pertussis; Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Haemophilus Infections | interventions — Tetanus Toxoid; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects in Study 494-01 and Study 494-03 who had received 4 doses of Pentacel™ vaccine.
  Interventions: Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis (DAPTACEL®)

INTERVENTIONS:
Biological: Diphtheria and Tetanus Toxoids and Acellular Pertussis (DAPTACEL®) — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®

SUMMARY:
Objectives:

* To present the rates of adverse reactions after a dose of DAPTACEL® vaccine administered to children 4 to 6 years of age who have previously received four doses of PENTACEL™ vaccine.
* To present immunogenicity before and after a single dose of DAPTACEL® vaccine administered to children 4 to 6 years of age who have previously received four doses of PENTACEL™ vaccine.

DETAILED DESCRIPTION:
This study is designed to assess the safety and immunogenicity of DAPTACEL® vaccine administered at 4 to 6 years of age according to the US standard of care. The study population consists of PENTACEL™-primed subjects from Aventis Pasteur's pivotal studies 494-01 and 494-03. These children will receive DAPTACEL® vaccine as a 5th dose immunization between 4 to 6 years of age.

ELIGIBILITY:
Inclusion Criteria :

* Aged ≥ 4 years and 6 years.
* Signed and dated Investigational Review Board-approved informed consent from a parent or legally authorized representative.
* Judged to be in good health on the basis of reported medical history and physical examination.
* Able and willing to attend the scheduled visits and to comply with the study procedures.
* Has documented complete infant series and 4th dose in Study 494-01 or Study 494-03, consisting of four previous administrations of PENTACEL™.

Exclusion Criteria :

* Received a 5th dose of DTaP-containing vaccine scheduled at 4 to 6 years of age.
* Serious underlying chronic disease, including, but not limited to:
* Diabetes mellitus; malignancy; cardiopulmonary disease; renal, endocrinologic, or hepatic dysfunction; or hematologic disorder; or
* Unstable or evolving neurologic disorders that may predispose the subject to seizures or neurologic deterioration.
* Known or suspected primary or acquired disease of the immune system.
* Administration of immune globulin or other blood products within the last 3 months, or injected or oral corticosteroids or other immunomodulatory therapy within 6 weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting <7 days may be included in the trial as long as they have not received more than 1 course within the last 2 weeks prior to enrollment.
* Had allergy shots started or had changes in regimen or dosing of allergy shots within the last 4 weeks.
* Receipt of any other vaccine within the past 30 days, or planning to receive another vaccine within 30 days before the Visit 2 blood draw, with the exclusion of M-M-R®II and IPV.
* Any other condition which, in the opinion of the Investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Enrolled in another vaccine trial.
* Personal history of physician-diagnosed or laboratory-confirmed pertussis disease within the past 30 months.
* Known or suspected allergy to any of the vaccines or vaccine components intended for use in this study.

Temporary contraindications:

* A subject who meets either of the following criteria at the time of planned vaccination will have enrollment deferred until complete resolution of symptoms:

Oral temperature ≥ 100.4°F (≥ 38.0ºC) (Note: A tympanic thermometer should not be used).

* Any moderate or severe acute illness with or without fever.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 989 (Actual)
Dates: Start 2004-02; Primary Completion 2005-06 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (19):
- United States (19):
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Oakland, California
  - Torrance, California
  - Orlando, Florida
  - Atlanta, Georgia
  - Boston, Massachusetts
  - Woburn, Massachusetts
  - Omaha, Nebraska
  - Albany, New York
  - Rochester, New York
  - Chapel Hill, North Carolina
  - Sylva, North Carolina
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - San Antonio, Texas
  - Layton, Utah
  - Vancouver, Washington
  - Marshfield, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 05 February through 30 November 2004 at 19 US sites.
Pre-assignment Details: A total of 989 participants were enrolled and vaccinated with DAPTACEL as the fifth dose after receiving 4 doses of Pentacel vaccine in previous studies.
Groups:
- DAPTACEL® Vaccine Group: Participants received DAPTACEL® as the 5th dose after 4 doses of Pentacel® in Study 494-01 or Study 494-03.
Period: Overall Study
Arm/Group | DAPTACEL® Vaccine Group
Started | 989
Completed | 976
Not Completed | 13
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 989
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 989
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.2 (0.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 514
  Male | 475
Region of Enrollment [Number; unit: participants]
  United States | 989

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Percentage of Participants With 4-Fold Rises in Anti-Pertussis Post-vaccination With DAPTACEL® as a Fifth Dose.
Description: Anti-pertussis (anti-Pertussis, anti-Filamentous Haemagglutinin, anti-Fimbriae, and anti-Pertactin).
  Fold-rise is calculated as Post-Dose 5/Pre-Dose 5 titer.
Time Frame: Day 28 to 48 Post-dose 5
Population: The vaccine antibody responses were evaluated in a subset of the per-protocol population for immunogenicity.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 228
Percentage of Participants
  Anti-Pertussis (EU/mL) ≥ 4-Fold Rise | 94
  Anti-Filamentous Haemagglutinin ≥ 4-Fold Rise | 91
  Anti-Fimbriae Types 2 and 3 ≥ 4-Fold Rise | 91
  Anti-Pertactin (EU/mL) ≥ 4-Fold Rise | 90

2. Other Pre Specified Outcome: Percentage of Participants With Anti-Pertussis Booster Response Post-vaccination With DAPTACEL® as a Fifth Dose
Description: Booster response calculation: If Pre-Dose 5 titer < 4x limit of quantitation (LOQ), a 4-fold rise of Post-dose 5/Pre-dose 5; If Pre-dose 5 titer ≥ 4x LOQ, a 2-fold rise of Post-dose 5/Pre-dose 5.
Time Frame: Day 28 to 48 Post-dose 5
Population: The anti-Pertussis Booster response was evaluated in a subset of the per-protocol population for immunogenicity.
Measure: Number; unit: Percentage of participants
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 228
Percentage of participants
  Anti-Pertussis (EU/mL) | 98
  Anti-Filamentous Haemagglutinin | 97
  Anti-Fimbriae Types 2 and 3 | 96
  Anti-Pertactin (EU/mL) | 95

3. Other Pre Specified Outcome: Percentage of Participants With Anti-Diphtheria and Anti-Tetanus Seroprotection Pre- and Post-vaccination With DAPTACEL® as a Fifth Dose
Description: Seroprotection is defined as a titer of ≥ 0.01 IU/mL for both Diphtheria and Tetanus before the fifth dose booster vaccination
Time Frame: Day 28 to 48 Post-dose 5
Population: The anti-Diphtheria and anti-Tetanus Toxoids Responses were evaluated in a subset of the per-protocol population for immunogenicity.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 228
Percentage of Participants
  Anti-Diphtheria (IU/mL) ≥0.01 Pre-dose 5 | 100
  Anti-Diphtheria (IU/mL) ≥0.1 Pre-dose 5 | 77
  Anti-Diphtheria (IU/mL) ≥1.0 Pre-dose 5 | 9
  Anti-Diphtheria (IU/mL) ≥0.1 Post-dose 5 | 100
  Anti-Diphtheria (IU/mL) ≥1.0 Post-dose 5 | 100
  Anti-Tetanus (IU/mL) ≥0.01 Pre-dose 5 | 100
  Anti-Tetanus (IU/mL) ≥0.1 Pre-dose 5 | 92
  Anti-Tetanus (IU/mL) ≥1.0 Pre-dose 5 | 13
  Anti-Tetanus (IU/mL) ≥0.1 Post-dose 5 | 100
  Anti-Tetanus (IU/mL) ≥1.0 Post-dose 5 | 96

4. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Anti-Pertussis, Anti-Diphtheria, and Anti-Tetanus Toxoids Pre- and Post-vaccination With DAPTACEL® as a Fifth Dose
Time Frame: Pre-dose 5 and Day 28 to 48 Post-dose 5
Population: The GMTs of anti-Pertussis, anti-Diphtheria, and anti-Tetanus Toxoids Responses were evaluated in a subset of the per-protocol population for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 228
Titers
  Anti-Pertussis (EU/mL) - Pre-dose 5 | 12.73 [10.85 to 14.94]
  Anti-Pertussis (EU/mL) - Post-dose 5 | 309.64 [276.16 to 347.18]
  Anti-Filamentous Haemagglutinin (EU/mL) Pre-dose 5 | 9.90 [8.49 to 11.55]
  Anti-Filamentous Haemagglutinin (EU/mL) Post-dose5 | 158.27 [144.26 to 173.63]
  Anti-Fimbriae Types 2 and 3 (EU/mL) Pre-dose 5 | 40.62 [35.13 to 46.98]
  Anti-Fimbriae Types 2 and 3 (EU/mL) Post-dose 5 | 659.28 [595.32 to 730.12]
  Anti-Pertactin (EU/mL) Pre-dose 5 | 10.36 [8.92 to 12.02]
  Anti-Pertactin (EU/mL) Post-dose 5 | 140.86 [122.24 to 162.31]
  Anti-Diphtheria (IU/mL) Pre-dose 5 | 0.25 [0.22 to 0.28]
  Anti-Diphtheria (IU/mL) Post-dose 5 | 18.98 [17.10 to 21.07]
  Anti-Tetanus (IU/mL) Pre-dose 5 | 0.38 [0.33 to 0.42]
  Anti-Tetanus (IU/mL) Post-dose 5 | 4.30 [3.86 to 4.79]

5. Primary Outcome: Percentage of Participants With Solicited Local or Systemic Reactions Post-vaccination With DAPTACEL® as the Fifth Dose After 4 Doses of Pentacel®
Description: Solicited local reactions: Redness, swelling, tenderness at injection site, change in limb circumference, and limb function.
  Systemic reactions: Fever (temperature), irritability, crying, lethargy, appetite decreased, vomiting, diarrhea, and rash.
Time Frame: 0 to 3 days post-dose 5 vaccination
Population: Safety analysis was on all enrolled and vaccinated participants intend-to-treat population.
Measure: Number; unit: Percentage of Participants
Arm/Group | DAPTACEL® Vaccine Group
Number analyzed (Participants) | 982
Percentage of Participants
  Any Solicited Systemic Reaction Post-dose 5 | 62
  Any Redness (> 5 mm) | 20
  Grade 3 Redness (> 50 mm) | 7
  Any Swelling (> 5 mm) | 12
  Grade 3 Swelling (> 50 mm) | 3
  Any Tenderness | 50
  Grade 3 Tenderness (Incapacitating) | 0
  Any Change in Limb Circumference (> 5 mm) | 29
  Grade 3 Change in Limb Circumference (> 40 mm) | 1
  Any Functional Impairment | 9
  Grade 3 Functional Impairment (Incapacitating) | 0
  Any Solicited Systemic Reaction Post-dose 5 | 37
  Any Fever (≥ 38 ºC) | 5
  Grade 3 Fever (> 39.5 ºC) | 0
  Any Irritability | 23
  Grade 3 Irritability (Incapacitating) | 1
  Any Crying | 7
  Grade 3 Crying (Incapacitating) | 0
  Any Lethargy | 13
  Grade 3 Lethargy (Incapacitating) | 0
  Any Anorexia | 11
  Grade 3 Anorexia (Skips 2 meals) | 1
  Any Vomiting | 3
  Grade 3 Vomiting (≥ 3 episodes) | 1
  Any Diarrhea | 4
  Grade 3 Diarrhea (> 5 diarrhea stools) | 0
  Rash Present | 5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months post-vaccination.
Arm/Group | DAPTACEL® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 10/989
Other Adverse Events (participants affected / at risk) | 49/989
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPTACEL® Vaccine Group (N=989)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis nos (Infections and infestations) | 1 (1)
Pneumonia nos (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Febrile convulsion (Nervous system disorders) | 1 (1)
Obstructive sleep apnoea syndrome (Nervous system disorders) | 1 (1)
Asthma nos (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPTACEL® Vaccine Group (N=989)
Upper respiratory tract infection NOS (Infections and infestations) | 49 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications